CLINICAL TRIAL: NCT05879055
Title: A Phase II Study to Evaluate the Efficacy, Safety and Pharmacokinetics of PM8002 Injection in Combination With Chemotherapy as Second Line Therapy in Unresectable Neuroendocrine Neoplasm
Brief Title: A Study of PM8002 in Combination With Chemotherapy in Patients With NEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-B009C-NEN-R
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Neuroendocrine Neoplasm
Keywords: Second line; NEC; G3 NET
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002+FOLFIRI (Experimental): Subjects will be administered with PM8002 plus FOLFIRI via intravenously (IV) Q2W until disease progression or intolerable toxicity for a maximum of 2 years.
  Interventions: Drug: PM8002; Drug: FOLFIRI

INTERVENTIONS:
Drug: PM8002 — IV infusion
Drug: FOLFIRI — IV infusion

SUMMARY:
PM8002 is a bispecific antibody targeting PD-L1 and VEGF. This study will evaluate the efficacy and safety of PM8002 in combination with FOLFIRI as second line treatment for neuroendocrine neoplasm (NEC and Ki-67≥55% G3 NET).

DETAILED DESCRIPTION:
This is a phase II, single arm study assessing the efficacy and safety of PM8002 in combination with FOLFIRI as second line treatment for neuroendocrine neoplasm (NEC and Ki-67≥55% G3 NET) who failed first-line platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form before any trial-related processes;
2. Aged ≥ 18 years;
3. Ki-67≥55% G3 NET and NEC were confirmed histologically or cytologically by pathological diagnosis in this study;
4. Subjects failed first-line platinum-based chemotherapy;
5. Adequate organ function;
6. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1;
7. Expected survival ≥ 12 weeks;
8. Had at least one measurable tumor lesion according to RECIST v1.1;

Exclusion Criteria:

1. History of severe allergic disease, severe drug allergy or have known allergy to any component of the study drugs;
2. Evidence and history of severe bleeding tendency;
3. History of severe cardiovascular diseases within 6 months;
4. Subjects should provide formalin-fixed-paraffin-embedded (FFPE) tumor samples during the screening period (up to 24 months);
5. Current presence of uncontrolled pleural, pericardial, and peritoneal effusions;
6. History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation;
7. History of alcohol abuse, psychotropic substance abuse or drug abuse;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome;
9. Pregnant or lactating women;
10. Other conditions considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Duration of response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first
Progression free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1)
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Principal Investigator — Chinese PLA General Hospital
Locations (13):
- China (13):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Province Cancer Hospital, Fuzhou, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Union Hospital Tongji Medical College of Hust, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Yunnan Cancer Hospital (The Third Affiliated Hospital of Kunming Medical University), Kunming, Yunnan
  - Chinese PLA General Hospital, Beijing
  - ZhongShan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations.
Time Frame: After the trial completed.
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.